CLINICAL TRIAL: NCT00057356
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging Pilot Study Evaluating the Efficacy and Safety of YM087 in Patients With Decompensated Chronic Heart Failure
Brief Title: Safety and Efficacy Study of YM087 (Conivaptan) in Patients With Acute Decompensated Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sr Manager Clinical Trials Registry, Astellas Pharma US, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 087-CL-071
Record Dates: First submitted 2003-03-31; First posted 2003-04-01 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; YM078
MeSH Terms: interventions — conivaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental): Low dose
  Interventions: Drug: conivaptan
- 3 (Experimental): Middle dose
  Interventions: Drug: conivaptan
- 4 (Experimental): High dose
  Interventions: Drug: conivaptan

INTERVENTIONS:
Drug: conivaptan — IV
  Other Names: Vaprisol; YM087
  Arms: 2; 3; 4
Drug: placebo — IV
  Arms: 1

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose ranging pilot study to examine the effects of conivaptan in patients with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients may be male or female age 18 years or older.
* Women must be post-menopausal or surgically sterile.
* Patients must have chronic heart failure of at least 2 months duration and be hospitalized for the treatment of worsening heart failure. The primary manifestation of worsening heart failure must be worsening dyspnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2002-11; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in respiratory Visual analog Scale (VAS) | 48 hours

SECONDARY OUTCOMES:
Change from baseline in global VAS | 48 hours
Total urine output vs. baseline | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (26):
- United States (26):
  - The Heart Center, P.C., Huntsville, Alabama
  - LA County/USC Medical Center, Los Angeles, California
  - San Joaquin Cardiology, Manteca, California
  - Apex Research Institute, Santa Ana, California
  - The Greater Fort Lauderdale Heart Group Research, Fort Lauderdale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - U. Miami, Jackson Mem'l Medical Center, Miami, Florida
  - Discovery Medical Research Group, Ocala, Florida
  - Rush-Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Louisiana State University Medical Center School of Medicine, New Orleans, Louisiana
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Cardiac Centers of Louisiana, LLC, Shreveport, Louisiana
  - University of Maryland Hospital, Baltimore, Maryland
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Presbyterian Hosp, Milstein Hosp., New York, New York
  - University of Cincinnati, College of Medicine, Div. of Cardiology, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Heart and Lung Research Institute, Columbus, Ohio
  - Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baptist Clinical Research, Memphis, Tennessee
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington